CLINICAL TRIAL: NCT02480530
Title: Evaluating Individual and Patient-Selected Family/Friend/or Reciprocal Peer Notifications to Improve Statin Medication Adherence Among Patients With Coronary Artery Disease
Brief Title: Using Feedback Reports to Improve Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 01461
Record Dates: First submitted 2014-05-01; First posted 2015-06-24 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease; Adherence
Keywords: Medication Adherence; Reciprocal Peer; Telemonitoring
MeSH Terms: conditions — Coronary Artery Disease; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Patients will be given educational material on the importance of adherence to statin medications. The GlowCaps device will be set to only record adherence.
- Individual Feedback (Experimental): In addition to educational material on adherence to statin medications, the research coordinator will review set-up of personal reminders for the GlowCaps device which will be set to glow and buzz when the medication is missed. In addition, patients will receive information on the weekly adherence feedback report.
  Interventions: Behavioral: Individual Feedback
- Feedback Friend (Experimental): The patient will be given educational material on the importance of adhering to statin medications. The research coordinator will review set-up of alarm features of GlowCaps device. Similar to Arm 2, patients will be given information on interpretation of weekly adherence feedback report. If the patient chooses a family/friend, they will be called and provided information on the interpretation of weekly adherence feedback report. If the patient chooses a reciprocal partner, they will be assigned to another patient who has made a similar choice
  Interventions: Behavioral: Individual Feedback; Behavioral: Feedback Friend

INTERVENTIONS:
Behavioral: Individual Feedback — Patient gets feedback reports on adherence weekly.
  Arms: Feedback Friend; Individual Feedback
Behavioral: Feedback Friend — In addition to individual feedback reports this information will be sent to an assigned family/friend or reciprocal peer.
  Arms: Feedback Friend

SUMMARY:
The purpose of this research study is to improve statin medication adherence among Veterans with coronary artery disease with poor adherence to medications. The investigators are testing if newer technology pill bottle devices linked with individual feedback and/or social incentive strategies can improve medication taking behavior.

DETAILED DESCRIPTION:
Patients with coronary artery disease and previous poor adherence to statin medications will be recruited at Philadelphia VA Medical Center. Enrolled participants will be randomly assigned to one of three arms:

1. Control Group
2. Individual Alarm device and feedback report
3. Individual plus patient-selected Feedback Friend report

Patients will be given a medication-monitoring device (Vitality GlowCaps) to monitor the statin medication that is being currently prescribed by their primary care physician. In first group, the control arm (Arm 1), the device reminders will be turned off but the device will continue recording adherence to the medications. In second group, reminder arm (Arm 2), the device will be programmed as an alarm that will be activated if the patient does not take the medication at the time set by the patient. In addition the patient will get a weekly report of his/her adherence. In the third group, patient-selected family/friend/or reciprocal peer feedback arm (Arm 3), in addition to the activation of the alarm function the device will be linked to a weekly report on adherence to medications. This report will be delivered to the patient and to the patient identified family/friend/ or reciprocal peer.

ELIGIBILITY:
Inclusion Criteria:

* All participants will have a diagnosis of CAD
* To be eligible they must be between the ages of 30-75 years of age-to ensure we are targeting those most likely to benefit from improving control to these medications
* Patients must have been prescribed a statin by their provider and a documented poor adherence as measured by a 16-month medication adherence rate (Medication Possession Ratio) of <80%

Exclusion Criteria:

* Due to the use of the medication adherence reminder device, patients must speak English
* Have a home address
* Telephone number
* Be willing and able to identify a friend or family member
* The investigators will exclude atients with active substance abuse, significant hearing loss, or reduced cognitive ability as determined from the patient's problem list

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09-03 (Actual); Study Completion 2015-09-03 (Actual)

PRIMARY OUTCOMES:
Adherence | Change in baseline adherence at 3 month and 6 month
  Adherence will be measured using the following formula: [Number of times the pill bottle was opened/(Number of times a day each medication is prescribed to be taken multiplied by the total number of days in study)].

SECONDARY OUTCOMES:
Patient Activation | Change in baseline patient activation at 3 month and 6 month
  The investigators will utilize the 13-item Patient Activation Measure (PAM) to measure an individual's activation level.18 This tool has been used in previous studies to predict self-efficacy for health behaviors, such as exercise and medications adherence. Response categories for each item are strongly agree, agree, disagree and strongly disagree. Responses are then scaled and transformed to a score ranging from 0 to 100. These scores are correlated with four stages of activation.
Social Support | Change in baseline social support at 3 month and 6 month
  The multidimensional scale of perceived social support will be given at baseline, 3-months, and 6-months. This is a 12-item questionnaire is a validated measure of social support. For each item, respondents must choose one answer that reflects their assessment of social support on a 7-point scale.19 The items divide into 3 main factors of support: Family, Friends, and Significant other.
LDL levels | Change in baseline LDL level at 6 month
  The investigators will obtain baseline LDL levels for each patient prior to the intervention. In addition to monitor impact of adherence to the statin medication the investigators will obtain LDL levels at baseline and 6-month time periods for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Reddy, MD, Principal Investigator — University of Pennsylvania/Philadelphia VAMC; Judith Long, MD, Principal Investigator — University of Pennsylvania Assistant Professor
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Reddy A, Huseman TL, Canamucio A, Marcus SC, Asch DA, Volpp K, Long JA. Patient and Partner Feedback Reports to Improve Statin Medication Adherence: A Randomized Control Trial. J Gen Intern Med. 2017 Mar;32(3):256-261. doi: 10.1007/s11606-016-3858-0. Epub 2016 Sep 9. PMID 27612487